CLINICAL TRIAL: NCT02597829
Title: Does Clinical Response Correlate With Serum Certolizumab Levels? A Prospective Open Label Trial of Adult Patients With Active Crohn's Disease (APOLLO)
Brief Title: Does Clinical Response Correlate With Serum Certolizumab Levels?
Acronym: APOLLO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shafran Gastroenterology Center (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ShafranGC
Record Dates: First submitted 2015-10-27; First posted 2015-11-05 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Crohn's Disease
Keywords: Inflammatory Bowel Disease; Mucosal Healing; Certolizumab pegol
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label Certolizumab Pegol (Other): Active Treatment
  Interventions: Drug: Certolizumab Pegol

INTERVENTIONS:
Drug: Certolizumab Pegol — Subcutaneous Injection
  Other Names: Cimzia

SUMMARY:
A prospective open label trial of adult patients with active Crohn's disease to determine if plasma concentrations of certolizumab pegol correlate to mucosal healing.

ELIGIBILITY:
Subject Inclusion Criteria

1. Males and females ≥ 18 and ≤ 70 years of age.
2. Diagnosis of colonic, ileocolonic, or ileal Crohn's disease for ≥ 3 months confirmed by radiography, histology, and/or endoscopy at any time in the past.
3. Moderately to severely active Crohn's disease as defined by a Harvey Bradshaw

   Index (HBI) ≥ 8 at baseline AND at least one of the following:
   * Abnormal CRP at screening (> Upper Limit of Normal [ULN] accepted lab assay)
   * Elevated fecal calprotectin at screening (> ULN accepted lab assay)
   * Endoscopic evidence (colonoscopy or small bowel video capsule endoscopy) of active Crohn's ulcerations within 3 months of baseline or during screening
4. Taking a stable dose of corticosteroids (oral or anorectal) ≤ 40 mg/day, or equivalent, for at least 2 weeks prior to baseline.
5. Taking a stable dose of 5-ASA, antibiotics, anti-diarrheals, analgesics, and/or probiotics for at least 4 weeks prior to baseline.
6. Taking a stable dose of immunosuppressants for at least 8 weeks prior to baseline.
7. Have screening laboratory test results within the following parameters:

   * Hemoglobin ≥ 8.5 g/dL
   * WBC count ≥ 3.5 x 103 µL
   * Neutrophils ≥ 1.5 x 103 µL
   * Platelets ≥ 100 x 103 µL
   * Serum creatinine < 1.7 mg/dL
   * AST and ALT concentrations must be within 2 times the ULN range for the laboratory conducting the test
8. Subject has a negative TB Screening Assessment (including a PPD test) and negative chest x-ray (posterior-anterior or PA and lateral view) within 2 months prior to screening.
9. If female, subject is either not of childbearing potential, defined as postmenopausal (> 45 years of age with amenorrhea for at least 18 months) or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, hysterectomy or otherwise incapable of pregnancy) or is of childbearing potential and is practicing on of the following methods of birth control:

   * Implants, injectables, some intrauterine devices (IUDs), intrauterine hormone releasing system (IUS), hormonal prescription oral contraceptives, contraceptive patch, or double barrier method
   * Male partner sterilization
   * Not heterosexually active
10. Negative serum pregnancy test at screening and a negative urine pregnancy test at baseline.
11. If male, not surgically sterile, and heterosexually active with a woman of child bearing potential, subject must agree to use a double barrier method of birth control and not donate sperm during the study and for 12 weeks after receiving study agent.
12. Subject must be able and willing to give written informed consent and to comply with the requirements of the study protocol.

Subject Exclusion Criteria

1. Any and all contraindications to the use of certolizumab pegol including: active or latent TB, active viral infection or chronic recurrent infections, evidence of dysplasia or history of malignancy, congestive heart failure (CHF), demyelinating disease and cytopenia.
2. Subject who previously received treatment with certolizumab pegol or previously participated in a certolizumab pegol study.
3. Has complications of Crohn's disease such as symptomatic strictures or stenoses, short bowel syndrome, or any other manifestation that might be anticipated to require surgery, could preclude the use of the HBI to assess response to therapy, or would possibly confound the ability to assess the effect of treatment with certolizumab pegol.
4. Subject has had surgical bowel resection(s) within 6 months or any other intra- abdominal surgery within 3 months prior to baseline.
5. Subject with an ostomy or ileoanal pouch.
6. Subject has received anti-TNF agents < 8 weeks prior to baseline.
7. Subject has received other immunomodulatory biologic agents, < 8 weeks or within 5 half-lives of agent prior to baseline, whichever is longer
8. Subject is known to be infected with HIV, Hepatitis B or Hepatitis C
9. Subject with positive Clostridium difficile (C. difficile) toxin stool assay during the Screening period.
10. Subject has severe, progressive or uncontrolled renal, hepatic, hematological, endocrine, pulmonary, cardiac, neurologic, cerebral, or psychiatric disease, or signs and symptoms
11. Has a known history or lymphoproliferative disease, including lymphoma, or signs and symptoms suggestive or possible lymphoproliferative disease, such as lymphadenopathy or splenomegaly
12. History of clinically significant drug or alcohol abuse in the 12 months prior to baseline.
13. Female subjects who are pregnant, breast-feeding, or planning to become pregnant or a man who plans to father a child while enrolled in this study or within 20 weeks after the last dose of study agent.
14. Subject is considered by the Investigator, for any reason, to be an unsuitable candidate for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-11; Primary Completion 2018-05 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who achieve endoscopic improvement. | 20 Weeks

SECONDARY OUTCOMES:
Proportion of subjects who achieve clinical response. | 20 Weeks
Proportion of subjects who achieve clinical remission. | 20 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ira Shafran, M.D., Principal Investigator — Shafran Gastroenterology Center
Locations (1):
- Shafran Gastroenterology Center, Winter Park, Florida, United States